CLINICAL TRIAL: NCT02964611
Title: Assessing Changes in Social Cognition and Personality in Patients with Frontotemporal Lobar Degeneration, Alzheimer's Disease and Parkinson's Disease and Their Effect on the Patient-caregiver Relationship
Brief Title: Social Cognition and Personality Changes in Alzheimer's & Parkinson's Disease & Frontotemporal Lobar Degeneration
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Carmela Tartaglia, Principal Investigator, University Health Network, Toronto
Other Study IDs: 12-0451-BE
Record Dates: First submitted 2016-09-23; First posted 2016-11-16 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer's Disease; Parkinson's Disease; Frontotemporal Lobar Degeneration
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Frontotemporal Lobar Degeneration | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Alzheimer's disease: Observational Study
  Interventions: Behavioral: Observational Study
- Parkinson's disease: Observational Study
  Interventions: Behavioral: Observational Study
- Frontotemporal Lobar Degeneration: Observational Study
  Interventions: Behavioral: Observational Study
- Healthy Controls: Observational Study
  Interventions: Behavioral: Observational Study

INTERVENTIONS:
Behavioral: Observational Study — This is an observational study.

SUMMARY:
The aim of this study is to compare personality and social cognition changes, including emotion detection and self-awareness, and neuroanatomical correlates in patients, and how that affects the caregiver-patient relationship.

DETAILED DESCRIPTION:
The purpose of this study is to understand social cognition changes in patients with Alzheimer's disease (AD), Parkinson's disease (PD), and Frontotemporal Lobar Degeneration (FTLD), which includes Progressive Supranuclear Palsy (PSP), Corticobasal Syndrome (CBS) and Frontotemporal Dementia (FTD - behavioural variant frontotemporal dementia, progressive non-fluent aphasia and semantic dementia), and the effect of these changes on the patients' relationship with their caregivers. In addition, the study aims to provide a greater clarity in the neuroanatomical correlates of social cognition in patients with FTLD, PD and AD.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* ability to speak and understand the English language (as questionnaires and tests are only available in English)

Caregivers:

* primary caregiver for a given patient
* ability to speak and understand the English language (as questionnaires and tests are only available in English)

Exclusion Criteria:

Patients and Caregivers:

* history of another neurological disorder
* psychiatric disorder
* severe aphasia (semantic word loss)
* visual deficits requiring correction beyond the use of eyeglasses or contact lenses (intact visual acuity is required for completing both the questionnaires and the emotion evaluation test which consists of video vignettes)
* auditory deficits requiring correction beyond hearing aids (videos have auditory component)

Patients:

* presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body will be excluded as they will be unable to have a MRI scan.
* premenopausal women will be excluded due to the unknown risk of MRIs during pregnancy.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Alzheimer's disease, Parkinson's disease or Frontotemporal Lobar Degeneration
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

PRIMARY OUTCOMES:
Personality via the Interpersonal Adjectives Scales and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses interpersonal aspects of personality
Personality via the Behaviour Inhibition/Approach Scale (BIS/BAS) and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses the behavioural approach system that regulates appetitive motives, in which the goal is to move toward something desired, and the behavioural avoidance (or inhibition) system that regulates aversive motives, in which the goal is to move away from something unpleasant
Personality via the Big Five Inventory (BFI) and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses the patient's Big Five dimensions (openness, conscientiousness, extraversion, agreeableness, and neuroticism) with respect to past and current behavior
Social cognition via Social Norms Questionnaire and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses the patient's understanding of culturally relevant social norms
Social cognition via Interpersonal Reactivity Index (IRI) and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses the patient's empathy or ability to share in another's mental and emotional experience
Social cognition via Revised Self-Monitoring Scale (RSMS) and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses the patient's sensitivity to the expressive behaviour of others and their ability to monitor their self-presentation
Social cognition via Social Behaviour Observer Checklist and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses behaviors specific to behavioural variant Frontotemporal Dementia (bvFTD) and is helpful in differentiating bvFTD versus Alzheimer's disease.
Neuropsychiatric Inventory (NPI) and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses 12 neuropsychiatric disturbances commonly encountered in patients with dementia, including: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behaviour, night-time behaviour disturbances, and appetite and eating abnormalities
Clinical Dementia Rating Scale (CDR) and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses 8 domains of global dementia, including: memory, orientation, judgment/problem solving, community affairs, home and hobbies, personal care, behavioural comportment and personality, and language
Functional Activities Questionnaire (FAQ) and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses functional capacity in older adults
Behavioural Tests composite score and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Orientation, Digit span backward and forward, Naming, Modified trails, Benson figure copy, Cerad, Clock draw
Emotion Evaluation Task (EET) portion of The Awareness of Social Inference Test and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses the recognition of six basic emotions commonly recognized across cultures (happiness, sadness, anger, surprise, disgust, fear) as well as a seventh "neutral" emotion. The emotions are presented via video vignettes. After viewing each scene, the patient will be asked to choose the emotion represented from a list of seven emotional categories. The caregiver will complete the test separately, and be asked both to guess the emotion in each vignette, and to speculate on which emotion the patient will guess.
Geriatric Depression Scale (GDS) and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Assesses mood and depression in geriatric patients
Neuroimaging and differences between AD, PD, and FTLD | one time visit, through study completion of 3 years
  Functional connectivity of networks associated with social cognition and personality

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Tartaglia, M.D., Principal Investigator — Toronto Western Hospital, UHN; Tanz CRND
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No